CLINICAL TRIAL: NCT00666159
Title: A Randomized, Investigator Blinded Study of Protopic (Tacrolimus) Ointment Vs. Elidel (Pimecrolimus) Cream in Pediatric Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Comparison Study Between Protopic (Tacrolimus Ointment) and Elidel (Pimecrolimus Cream) in Treating Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-02-005
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; Protopic; Pediatric
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus; pimecrolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment
- 2 (Active Comparator)
  Interventions: Drug: pimecrolimus cream

INTERVENTIONS:
Drug: tacrolimus ointment — topical
  Other Names: Protopic; FK506 ointment
  Arms: 1
Drug: pimecrolimus cream — topical
  Other Names: Elidel
  Arms: 2

SUMMARY:
Comparison of Protopic Ointment to Elidel Cream to assess the safety and efficacy in pediatric patients with Atopic Dermatitis

DETAILED DESCRIPTION:
This is a two arm, randomized, investigator blinded study to compare Protopic Ointment to Elidel Cream in treating pediatric patients with moderate to severe Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Atopic Dermatitis which is rated moderate, severe or very severe using the Investigator's Global Atopic Dermatitis Assessment involving a minimum of 5% of the body's surface area
* If female, and of childbearing potential, patient has a negative pregnancy test and agrees to practice effective birth control during the study

Exclusion Criteria:

* Patient has a skin disorder other than Atopic Dermatitis in the areas to be treated
* Patient has extensive scarring or pigmented lesions in the areas to be treated that would interfere with rating of efficacy parameters
* Patient has clinically infected Atopic Dermatitis at baseline
* Patient is likely to require systemic corticosteroids, or the patient is likely to require intranasal or inhaled corticosteroids for an off-label indication or at higher doses than the maximum labeled dosing for the drug
* Patient has a known hypersensitivity to macrolides or any excipient of either study medication
* Patient has a chronic condition which is either not stable or not well controlled
* Patient is pregnant or breast feeding an infant

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2002-12; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Change Eczema Area and Severity Index (EASI) | 6 Weeks

SECONDARY OUTCOMES:
Investigator's Global Atopic Dermatitis Assessment (IGADA) | 6 Weeks
Patient's evaluation of itch | 6 Weeks
Body surface area affected | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Director — Astellas Pharma US, Inc.
Locations (11):
- United States (11):
  - New Haven, Connecticut
  - Miami, Florida
  - Chicago, Illinois
  - Boston, Massachusetts
  - Clinton Township, Michigan
  - Omaha, Nebraska
  - Reno, Nevada
  - Chapel Hill, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Houston, Texas

REFERENCES:
- [Background] Paller AS, Lebwohl M, Fleischer AB Jr, Antaya R, Langley RG, Kirsner RS, Blum RR, Rico MJ, Jaracz E, Crowe A, Linowski GJ; US/Canada Tacrolimus Ointment Study Group. Tacrolimus ointment is more effective than pimecrolimus cream with a similar safety profile in the treatment of atopic dermatitis: results from 3 randomized, comparative studies. J Am Acad Dermatol. 2005 May;52(5):810-22. doi: 10.1016/j.jaad.2004.12.038. PMID 15858471
- [Background] Kirsner RS, Heffernan MP, Antaya R. Safety and efficacy of tacrolimus ointment versus pimecrolimus cream in the treatment of patients with atopic dermatitis previously treated with corticosteroids. Acta Derm Venereol. 2010;90(1):58-64. doi: 10.2340/00015555-0748. PMID 20107727